CLINICAL TRIAL: NCT06614985
Title: The Efficacy and Safety of Treatment With Telitacicept in Primary Membranous Nephropathy
Acronym: TEST-T-PMN
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Huiming Wang, Director, Department of Nephrology, Renmin Hospital of Wuhan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Huiming Wang
Record Dates: First submitted 2024-05-30; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — telitacicept; Prednisone; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: After completing the induction treatment period, patients undergo an efficacy evaluation to determine if complete remission or partial remission has been achieved. Patients who have not achieved complete or partial remission are classified as non-responders. Patients who have achieved complete or partial remission are then randomly assigned to either Group A or Group B at a 1:1 ratio. Non-responders are also randomly assigned to either Group C or Group D at a 1:1 ratio. Treatment administration is subsequently carried out based on group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Active Comparator): After completing the induction treatment period, patients undergo an efficacy evaluation to determine if complete remission or partial remission has been achieved. Patients who have not achieved complete or partial remission are classified as non-responders. Patients who have achieved complete or partial remission are then randomly assigned to either Group A or Group B at a 1:1 ratio.
  Medication regimen of Group A： Prednisone：the maintenance induction treatment regimen is continued, with regular tapering (reducing by 5 mg every 2 weeks) until discontinuation； Cyclophosphamide injection：an intravenous injection of 0.4 g is administered twice a month.
  Interventions: Drug: Prednisone; Drug: Cyclophosphamide
- Group B (Experimental): Medication regimen of Group B： Prednisone：the maintenance induction treatment regimen is continued, with regular tapering (reducing by 5 mg every 2 weeks) until discontinuation； Telitacicept injection：an intravenous injection of 0.4 g is administered twice a month.
  Interventions: Drug: Telitacicept; Drug: Prednisone
- Group C (Active Comparator): After completing the induction treatment period, patients undergo an efficacy evaluation to determine if complete remission or partial remission has been achieved. Patients who have not achieved complete or partial remission are classified as non-responders. Non-responders are randomly assigned to either Group C or Group D at a 1:1 ratio.
  Medication regimen of Group C： Prednisone：the maintenance induction treatment regimen is continued, with regular tapering (reducing by 5 mg every 2 weeks) until discontinuation； Cyclophosphamide injection：an intravenous injection of 0.4 g is administered twice a month.
  Interventions: Drug: Prednisone; Drug: Cyclophosphamide
- Group D (Experimental): Medication regimen of Group D： Prednisone：the maintenance induction treatment regimen is continued, with regular tapering (reducing by 5 mg every 2 weeks) until discontinuation； Telitacicept injection：an intravenous injection of 0.4 g is administered twice a month.
  Interventions: Drug: Telitacicept; Drug: Prednisone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Telitacicept — Subcutaneous injection of 160 mg is administered once a week.
  Arms: Group B; Group D
Drug: Prednisone — Induction therapy period (3 months)：Eligible subjects receive induction treatment with Methylprednisone 0.5 g i. v. for 3 consecutive day and followed by orally administration of prednisone at an initial dose of 0.8 mg/kg/day, tapered gradually after 2 months (reduced by 5 mg every 2 weeks) Grouped treatment period (6 months): The maintenance induction treatment regimen is continued, with regular tapering (reducing by 5 mg every 2 weeks) until discontinuation.
Drug: Cyclophosphamide — An intravenous injection of 0.4 g is administered twice a month.
  Arms: Group A; Group C; Group D

SUMMARY:
This is a multiple-center, prospective, open-label, positive drug controlled, randomized, clinical study to evaluate the safety and efficacy of Telitacicept in the treatment of primary membranous nephropathy.

DETAILED DESCRIPTION:
The study consists of four stages as follows:

1. Screening period (0-6 months): After signing the informed consent form, subjects enter the screening period.
2. Induction treatment period (3 months): Eligible subjects receive induction treatment with Methylprednisone 0.5 g i. v. for 3 consecutive day and followed by orally administration of prednisone at an initial dose of 0.8 mg/kg/day, tapered gradually after 2 months (reduced by 5 mg every 2 weeks), and cyclophosphamide is administrated intravenously at a dose of 0.4 g/d twice a month.
3. Group treatment period (6 months): Patients who complete the induction treatment period undergo an efficacy assessment to determine whether they achieve a complete remission or partial remission. Patients who do not achieve a complete remission or partial remission are defined as non-responders. Patients who achieve a complete remission or partial remission are randomized and enter the group A or group B. Patients of non-responders are randomized and enter the group C and group D. Patients in group A and C continue the initial treatment regimen for 6 months. Patients in group B and D commence hypodermic injection of Telitacicept 160 mg weekly 6 months with the continued administration of prednisone and cyclophosphamide in group D while discontinued cyclophosphamide administration in group B.
4. Follow-up period (12 months): After completing 6 months of group treatment, cyclophosphamide or Telitacicept is discontinued with minimal dose of 5mg/d prednisone remained. All the patients are subjected to a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of primary membranous nephropathy through renal biopsy to be eligible for inclusion in the study.
2. Adult patients aged 18 years or older of any gender are eligible for inclusion in the study.
3. Patients who meet the diagnostic criteria for nephrotic syndrome, which includes quantitative urine protein levels greater than 3.5 g/24 h and serum albumin levels less than 30 g/L, are eligible for inclusion in the study.
4. Patients who meet the high-risk criteria for progression of membranous nephropathy based on the KDIGO (Kidney Disease: Improving Global Outcomes) guidelines are eligible for inclusion in the study. High-risk criteria include eGFR less than 60 mL/min/1.73 m2 and/or urine protein excretion greater than 8 g/day for at least 6 months, or normal eGFR with urine protein excretion greater than 3.5 g/day and urine protein reduction less than 50% after 6 months of ACEI/ARB treatment, with any of the following criteria: serum albumin less than 25 g/L, anti-PLA2R antibody greater than 50 RU/mL, urine α1-microglobulin greater than 40 μg/min, urine IgG1 greater than 1 μg/min, urine β2-microglobulin greater than 250 mg/day, and SI greater than 0.2.
5. Participants are required to consent to use effective contraception methods with their partners throughout the entire duration of the study. Participants must have a thorough understanding of the nature, significance, potential benefits, inconveniences, and potential risks of the study and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Secondary membranous nephropathy patients (caused by autoimmune or infectious diseases, tumors, etc.);
2. Patients with HIV infection, viral hepatitis, active liver disease (with ALT/AST/bilirubin levels exceeding 3 times the upper limit of normal), or other severe infections;
3. Patients with a rapid decline in eGFR (>15 mL/min) during the screening period are excluded;
4. Patients who have undergone kidney transplantation or other organ transplantation;
5. Patients with a known allergy or hypersensitivity to the active ingredient of the investigational drug or any of the listed excipients;
6. Patients with acute or critical cardiovascular or cerebrovascular diseases;
7. Patients with immunodeficiency, hypoalbuminemia (IgG < 400 mg/dl), or IgA deficiency (IgA < 10 mg/dL);
8. Pregnant or lactating women;
9. Patients diagnosed with malignant tumors within the past 5 years;
10. Laboratory findings of severe abnormalities (Hb < 80 g/L, PLT < 50,000/mm3, neutrophil count < 1,000/mm3, etc.);
11. Patients who have used steroids or immunosuppressive agents (including but not limited to corticosteroids, adrenocorticotropic hormones, azathioprine, mycophenolate mofetil, cyclophosphamide, methotrexate, leflunomide, tacrolimus, cyclosporine, biologic agents such as rituximab, etc.), cyclophosphamide, bortezomib, dexamethasone, Chinese medicines or preparations containing Tripterygium wilfordii, intravenous immunoglobulin, plasma exchange, leukapheresis, live vaccines, or other investigational drugs, etc., within 3 months prior to screening;
12. Patients with other diseases or conditions that, in the opinion of the investigator, would render the patient unsuitable for participation in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2024-10-20 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate at the end of follow-up (21 months post-treatment) | 21 months
  Complete remission defined as 24h urine protein quantification ≤0.3g/24h.
Partial remission rate at the end of follow-up (21 months post-treatment) | 21 months
  Partial remission defined as 24h proteinuria quantification <3.5g/24h or ≥50% reduction from baseline and stable serum creatinine or <30% increase from baseline value.

SECONDARY OUTCOMES:
Incidence of relapse of nephrotic syndrome at months 3, 6, 9, 12, 15, 18, and 21 after treatment | 3-21 months
  Recurrence of proteinuria >3.5 g/24h or at least a ≥50% increase from the nadir was defined as recurrence of nephrotic syndrome in patients who had achieved partial or complete remission.
Incidence of adverse events in each group | 0-21 months
  This trial specifies that the recording of adverse events shall be recorded as a medical history from the time the subject receives the induction phase treatment administration, and from the time of signing the informed consent form until the clinical diagnosis, abnormal signs and symptoms, and examination findings occurring prior to the administration of the induction phase treatment.
Complete remission rate at months 3, 6, 9, 12, 15, 18, and 21 after treatment | 3-21 months
  Complete remission defined as 24h urine protein quantification ≤0.3g/24h.
Partial remission rate at months 3, 6, 9, 12, 15, 18, and 21 after treatment | 3-21 months
  Partial remission defined as 24h proteinuria quantification <3.5g/24h or ≥50% reduction from baseline and stable serum creatinine or <30% increase from baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan university, Wuhan, Hubei China, China

IPD SHARING:
Plan to Share IPD: Undecided